CLINICAL TRIAL: NCT03279523
Title: F 18 T807 Tau PET Imaging of Older (>= 40 Years Old) HIV Infected (HIV+) and HIV Uninfected (HIV-) Individuals (IND 123119, Protocol G)
Brief Title: F 18 T807 PET (Positron Emission Tomograph )Scan for HIV Infected & Uninfected
Status: Completed | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IND 123119 Protocol G
Record Dates: First submitted 2016-05-03; First posted 2017-09-12 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease; HIV
Keywords: Dementia; HIV; Brain Disease; CNS Diseases; Mild Cognitive Impairment; Neurodegenerative Disease; Tauopathies
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Cognitive Dysfunction; Neurodegenerative Diseases; Tauopathies | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- F 18 T807: Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Interventions: Drug: F 18 T807

INTERVENTIONS:
Drug: F 18 T807 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: 18F-AV-1451

SUMMARY:
This project will collect quantitative pilot data that will allow the characterization of uptake and binding of 18F-AV-1451 (also known as F 18 T807, also known as T807, also known as 7-(6-fluoropyridin-3-yl)-5H-pyrido[4,3-b]indole), a novel tau imaging compound, in older HIV+ individuals with and without HAND and matched HIV uninfected (HIV-) controls. The primary goal is to develop this highly promising tau imaging technique as an biomarker of cognitive decline in HIV+ individuals. The investigators will obtain preliminary data that will support the possibility of detecting early brain pathological changes due to HIV. Data generated from this study will be used for submission of National Institutes of Health (NIH) grants comparing tau deposition in HAND compared to other neurodegenerative disorders. It is hypothesized that specific topographies will help distinguish these neurodegenerative disorders in older individuals.

DETAILED DESCRIPTION:
This protocol will demonstrate the presence of tau fibrils in older HIV+ patients with HIV associated neurocognitive disorders (HAND) compared to cognitively normal HIV+ individuals and HIV- controls.

It will also demonstrate that the phenoconversion from cognitively normal (CN) status to HAND will be closely correlated with neocortical F 18 T807 uptake. In particular, HIV+ patients with MND will have greater tau cortical deposition compared to ANI individuals.

The investigtors hypothesize that in vivo tau imaging will ultimately:

* Demonstrate the presence of tau fibrils in older HIV+ patients with HIV associated neurocognitive disorders (HAND) compared to cognitively normal HIV+ individuals and HIV- controls.
* Demonstrate that the phenoconversion from cognitively normal (CN) status to HAND will be closely correlated with neocortical F 18 T807 uptake. In particular, HIV+ patients with MND will have greater tau cortical deposition compared to ANI individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, ≥ 40 years of age.
2. Testing for HIV status. If positive will be included in the HIV+ group and if negative will be included in the HIV- group.
3. Females without documented history of menopause or hysterectomy will undergo a urine pregnancy test 24 hours prior to F 18 T807 drug administration.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severe chronic back pain might not be able to lie still during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a high risk for Torsades de Pointes or is taking medications known to prolong QT interval.
4. Has hypersensitivity to F 18 T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Currently pregnant or breast-feeding.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 HIV+ and 40 HIV- participants will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Perform human in vivo tau imaging using F 18 T807 in 30 older (≥ 40 years old) HIV+ participants and 30 HIV- controls. | 5 years

SECONDARY OUTCOMES:
: Correlate regional quantitative T807 binding potentials (BPs) with cognitive impairment, as documented by neuropsychological performance tests, in HIV+ and HIV- individuals. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of this study, we are obtaining data from the participant. We would like to use this data' for studies going on right now as well as studies that are conducted in the future. These studies may provide additional information that will be helpful in understanding cognitive impairment, or other diseases or conditions, including research to develop investigational tests, treatments, drugs or devices that are not yet approved by the U.S. Food and Drug Administration. It is unlikely that what we learn from these studies will have a direct benefit to the participant.